CLINICAL TRIAL: NCT06833749
Title: A Double-blind, Placebo-controlled, Randomized Study to Evaluate the Efficacy and Safety of KBP-336 As an Adjunct to Diet and Exercise in Obese Individuals with Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of KBP-336 in Obese Individuals with Osteoarthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: KeyBioscience AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KBP-336-CD-003; 2024-517264-27-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-05; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis in the Knee; Obesity
Keywords: Obesity; Osteoarthritis; KBP-336; Pain; Phase 2
MeSH Terms: conditions — Obesity; Osteoarthritis; Pain

STUDY DESIGN:
Intervention Model Description: Double-blind, Randomized, Placebo-controlled trial design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- KBP-336 Dose 1 (Active Comparator)
  Interventions: Drug: KBP-336
- KBP-336 Dose 2 (Active Comparator)
  Interventions: Drug: KBP-336
- KBP-336 Dose 3 (Active Comparator)
  Interventions: Drug: KBP-336

INTERVENTIONS:
Drug: KBP-336 — KBP-336 is a long acting Dual Amylin and Calcitonin Receptor agonist designed for weekly administration through subcutaneous injection.
  Arms: KBP-336 Dose 1; KBP-336 Dose 2; KBP-336 Dose 3
Drug: Placebo — Placebo to match KBP-336
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if KBP-336 works to treat pain in osteoarthritis in individuals living with obesity. It will also learn about the effects on other parameters, such as quality of life and metabolism, as well as safety of KBP-336. The main questions it aims to answer are:

* Does KBP-336 lower knee pain from osteoarthritis in individuals with obesity
* Does KBP-336 lower bodyweight in the same population. Researchers will compare KBP-336 to a placebo (a look-alike substance that contains no drug) to see if KBP-336 works to pain and obesity

Participants will:

* Take KBP-336 or a placebo every week for 6 months
* Visit the clinic once every 2 weeks for checkups and tests
* Keep a diary of their symptoms and the amount of medication they use in addition to KBP-336

ELIGIBILITY:
Inclusion Criteria:

1. The participant is able to read and understand the language and content of the study material and provide written Informed Consent.
2. Willing and able to comply with study requirements and instructions
3. A diagnosis of OA of the target knee based on American College of Rheumatology (ACR) clinical and radiographic criteria(31), with OA symptoms (as reported by the participant) that have been present for at least 3 months prior to screening
4. Radiological OA grade 2 or 3 of the target knee, using the Kellgren-Lawrence method as graded by a central reader on a Fixed-Flexion X-ray obtained during screening, or on a recent (within 6 months) X-ray which fulfills the protocol specifications for reading
5. Age ≥ 45 years of either sex
6. Body Mass Index (BMI) ≥ 30 kg/m2
7. Good health, defined as no significantly relevant medical history or findings on physical examination, vital signs, ECG, and laboratory results in the opinion of the investigator.
8. Intolerance or insufficient pain relief with standard of care (e.g. physiotherapy, paracetamol, local or systemic NSAID, short term opioid use, injections of hyaluronic acid, or corticosteroids) for symptomatic OA in the index knee in the opinion of the investigator.
9. WOMAC pain subscale score in target knee at screening AND baseline ≥20 (0-50 scale)
10. Willing to withdraw from any pain medication including, but not limited to, Opioids (including semisynthetic opioids), Non-Steroidal Anti-inflammatories (NSAIDs, with the exception of low-dose aspirin for thromboprophylaxis), COX-2 inhibitors, Topical medication, and Serotonin and Noradrenaline Reuptake Inhibitors (SNRIs e.g. Duloxetine) and only use the allowed Rescue Medications from baseline to Visit 13/ET (maximum 4000 mg paracetamol per day)

Exclusion Criteria:

1. Partial or complete joint replacement of either knee
2. Target knee surgery or arthroscopy within 1 year prior to screening
3. Diagnosis of OA resulting from trauma within the last 5 years
4. Pain of the contralateral knee exceeding that of the target knee at the baseline visit, as measured by the WOMAC pain subscale
5. Planned major surgery within the next 6 months
6. Uncontrolled thyroid disease in the opinion of the Investigator based on medical history and laboratory results collected in screening
7. Participant-reported weight loss >5% of body weight within the last 6 months of the screening visit
8. Bariatric surgery within the last 12 months of the screening visit
9. Current comorbid condition, other than OA, affecting target knee or systemic illness known to be significantly associated with arthritis or joint pathology affecting any joint, including but not necessarily limited to endocrinopathies, inflammatory, or autoimmune disease with significant joint involvement (e.g., Rheumatoid Arthritis); Seronegative Spondyloarthropathies (e.g. Ankylosing Spondylitis, Psoriasis arthritis, Reactive arthritis)
10. Conditions significantly affecting joint and bone health, in the opinion of the Investigator should be excluded (including but not limited to atrophic or hypotrophic OA, subchondral insufficiency fracture, osteonecrosis, osteoporotic fractures, excessive malalignment of the knee or severe chondrocalcinosis)
11. Active comorbid condition other than OA (e.g radicular back pain, bursitis, tendinitis) significantly affecting target knee pain reporting in the opinion of the investigator.
12. A Patient Health Questionnaire-9 (PHQ-9) score of ≥ 15 at screening
13. History of gout, or pseudogout, with high likelihood of flare up during trial participation that would require NSAID treatment, in the opinion of the investigator
14. Hip dislocation and congenital hip dysplasia with degenerative joint disease should be excluded.
15. Participation in any previous DACRA/amylin study
16. History or presence of clinically significant neurological disease or psychiatric disorder in the opinion of the investigator
17. Intra-articular injection of corticosteroids within 3 months or hyaluronic acid within 6 months of screening in the target knee or into any other major joint within 30 days prior to screening (for extended-release corticosteroid injections: within 6 months in target knee and 3 months into any other major joint).
18. Systemic corticosteroid treatment for the treatment of musculoskeletal conditions of more than 14 days during the past 6 months prior to screening.
19. Any pharmacological or non-pharmacological treatment primarily targeting OA started or changed during the 4 weeks prior to randomization or likely to be changed during the duration of the study
20. Treatment with medication for obesity, including GLP-1 analogues, unless the dose of use has been stable for at least six months prior to screening
21. Vitamin D deficiency defined as blood 25-OH D3 concentration ≤25 nmol/L. Vitamin D supplementation and subsequent rescreening is allowed
22. Presence or history of clinically significant allergies, including relevant drug hypersensitivity or allergy
23. Current malignancy or treatment for malignancy within the past five years, apart from resected basal cell carcinoma, squamous skin cell carcinoma, or resected cervical atypia or carcinoma in situ, unless affecting the target knee area.
24. History of alcohol or drug abuse within 5 years prior to screening, in the opinion of the Investigator.
25. Use of an investigational drug within 90 days prior to screening
26. For women of childbearing potential:

    1. Pregnancy (i.e. positive serum pregnancy test at screening) or breastfeeding
    2. Failure to agree to practice a highly effective method of contraception (see Appendix 2), from enrolment up to at least 3 months after the study end
27. For sexually active men with a female partner of childbearing potential:

    1. Failure to agree to ensure that their female partners use a highly effective method of contraception (see Appendix 2) from enrolment up to at least 3 months after the study end
    2. Failure to agree not to donate sperm throughout the study and at least 3 months after the study end
28. Unsuitable for study participation for any reason in the opinion of the Investigator.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The proportional change in body weight from baseline to endpoint | 183 Days
The change in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain scale from baseline to endpoint | 183 Days
  Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Following assessment the scores are normalized.

SECONDARY OUTCOMES:
Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) stiffness and function scales during the trial and at Day 183 | 183 Days
  Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Following assessment the scores are normalized.
Proportion of subjects reaching ≥5, ≥10 or ≥15% weight loss from baseline at Day 183 | 183 Days
Proportion of subjects reaching ≥30 and ≥50% reduction in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain scale from baseline at Day 183 | 183 Days
  Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Following assessment the scores are normalized.
Change from baseline in Assessment of Quality of Life 8 Dimensions (AQol 8D) at Day 183 | 183 Days
  The AQoL-8D consists of eight dimensions measured by 35 items with four to six levels each. Five out of eight dimensions assess the psychosocial domains of health: happiness, coping, self-worth, relationships, and mental health. The scale if from 0 - 1 and is calculated using (https://www.aqol.com.au/index.php/scoring-algorithms)
Change from baseline in Assessment of Quality of Life 8 Dimensions (AQol 8D) subscore Independent living at Day 183 | 183 Days
  The AQoL-8D consists of eight dimensions measured by 35 items with four to six levels each. Five out of eight dimensions assess the psychosocial domains of health: happiness, coping, self-worth, relationships, and mental health. The scale if from 0 - 1 and is calculated using (https://www.aqol.com.au/index.php/scoring-algorithms)
Change from baseline in the weekly average of daily pain using the Numerical Rating Scale (NRS) during the trial, and at Day 183 | 183 Days
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Area under the curve from baseline in the weekly average of daily pain using the Numerical Rating Scale (NRS) to Day 183 | 183 Days
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Change from baseline to Day 183 in waist-to-hip ratio | 183 Days
Change from baseline in whole body composition by DXA at Day 183 | 183 Days
Change from baseline in bone mineral density of the lumber spine, femoral head, and total hip by DXA at Day 183 | 183 Days
Change from baseline in Patient Global Assessment at Day 183 | 183 Days
Outcome Measures in Rheumatology (OMERACT) - Osteoarthritis Research Society International (OARSI) responder rates at Day 183 | 183 Days
Average weekly days using rescue medication | 183 Days

CONTACTS AND LOCATIONS:
Locations (20):
- Czechia (6):
  - Pratia Brno, s.r.o, Brno
  - L.K.N. Artrocentrum, Hlučín
  - Medical Plus, s.r.o, Hradiště
  - Pratia Pardubice a.s., Pardubice
  - Affidea Praha s.r.o, Prague
  - Pratia Prague, s.r.o, Prague
- Denmark (3):
  - Sanos Clinic Nordjylland, Gandrup
  - Sanos Clinic Herlev, Herlev
  - Sanos Clinic Syddanmark, Vejle
- Hong Kong Center for Clinical Research, Hong Kong, Hong Kong
- Moldova (3):
  - IMSP Sptalul Clinic Municipal "Sfanta Treime", Chisinau
  - PMSI Cardiology Institute/RTL SM SRL, Chisinau
  - Timofei Mosneaga Republican Clinical Hospital, Chisinau
- Poland (5):
  - NZOZ Bif-Med. s.c., Bytom
  - Medyczne Centrum Hetmańska, Poznan
  - DC-MED SP z o.o., Swidnica
  - NZOZ Lecznica MAK-MED s.c., Warsaw
  - Migre Polskie Centrum Leczenia Migreny, Wroclaw
- Romania (2):
  - Policlinica CCBR, Bucharest
  - Quantum Medical Bucharest, Bucharest

IPD SHARING:
Plan to Share IPD: No